CLINICAL TRIAL: NCT00607113
Title: Exploratory Study of Avastin (Bevacizumab) and RAD001 (Everolimus) in Advanced Low or Intermediate Grade Neuroendocrine Carcinoma (AVF3961s) (CRAD001C2481)
Brief Title: Avastin (Bevacizumab) and RAD001 (Everolimus) in Advanced Low or Intermediate Grade Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0954
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-05

CONDITIONS: Neuroendocrine Carcinoma
Keywords: Neuroendocrine Carcinoma; Avastin; Bevacizumab; RAD001; Everolimus
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Avastin (Experimental): Cycle 1 (First 3 weeks of study) - Avastin 15 mg/kg intravenous (IV)
  Interventions: Drug: Avastin
- Avastin + RAD001 (Experimental): Cycle 2: Avastin 15 mg/kg intravenous (IV) every 3 weeks + RAD001 10 mg orally daily for 3 weeks
  Interventions: Drug: Avastin; Drug: RAD001
- RAD001 (Experimental): Cycle 1 (First 3 weeks of study)- RAD001 10 mg orally daily for 21 Days
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: Avastin — 15 mg/kg By Vein Over 90 Minutes Every 21 Days
  Other Names: Bevacizumab
  Arms: Avastin; Avastin + RAD001
Drug: RAD001 — 10 mg By Mouth Daily For 21 Days
  Other Names: Everolimus
  Arms: Avastin + RAD001; RAD001

SUMMARY:
Primary Objectives:

* To determine the effect of Avastin on tumor blood flow as determined by functional computed tomography (CT) in patients with low or intermediate grade neuroendocrine carcinoma.
* To determine the effect of RAD001 on tumor blood flow as determined by functional CT in patients with low or intermediate grade neuroendocrine carcinoma.
* To determine the effect of adding the second agent (Avastin or RAD001) to the first agent (RAD001 or Avastin) on tumor blood flow as determined by functional CT

Secondary Objectives:

* To determine the clinical activity (objective response rate and progression free survival duration) of Avastin and RAD001 in patients with low or intermediate grade neuroendocrine carcinoma.
* To determine the biochemical response rate of Avastin and RAD001 in patients with low or intermediate grade neuroendocrine carcinoma.
* To determine the safety and tolerability of Avastin and RAD001 in patients with low or intermediate grade neuroendocrine carcinoma.

DETAILED DESCRIPTION:
The Study Drugs:

Avastin is designed to prevent the formation of new blood vessels that help cancer cells to grow. RAD001 is designed to block a protein that is important in the growth of cancer cells.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups. During Cycle 1, one group will receive Avastin and the other group will receive RAD001. Each study cycle is 3 weeks long. In Cycle 2 and every cycle after that, participants in both groups will receive both study drugs. There is an equal chance of being assigned to either group.

RAD001 Administration:

RAD001 tablets are taken once a day by mouth, followed by a large glass of water. The tablets are in a blister-pack under aluminum foil. The blisters should only be opened at the time you take the study drug.

You may either take RAD001 on an empty stomach or after a low-fat meal. Some examples of low-fat meals include: cereal with fat-free milk, muffin or bagel with fat-free spread, or fruit salad. You should avoid taking RAD001 after large fatty meals because this will lower the amount of RAD001 your body absorbs. Your dietary habits around the time you take RAD001 should be as consistent as possible throughout the study.

You should take RAD001 at about the same time each day. The study staff will give you a medication diary that you should bring to every study visit. You will be asked to use the diary by writing down the date and time you take RAD001, how many tablets you take, and any side effects you may experience.

Avastin Administration:

Avastin is given through a needle in a vein in the arm. The first dose will be given over about 90 minutes. If no intolerable side effects occur, the second dose will be given over about 60 minutes, and if again no intolerable side effects occur, each dose after that will be given over about 30 minutes.

Other Medications:

If you experience side effects from an Avastin infusion (such as fever/chills), you may receive additional medicine(s) at that time and before each later Avastin dose, in order to decrease the risk of side effects.

Study Visits:

On Day 1 of Cycle 1, you will receive your assigned study drug.

At the beginning of Cycle 2 and every cycle after that, you will be asked about any side effects you are experiencing. You will have a complete physical exam performed, including measurement of your vital signs and weight. Blood (about 3 teaspoons) and urine will also be collected for routine tests.

On Day 8 of Cycles 1 and 2 only, about 2 teaspoons of blood will be drawn for routine tests. These blood draws may be done at a local lab closer to your home.

Every 9 weeks, to check the status of the disease, you will have either CT scans or MRI scans of the tumor(s). The scans will be the same type that you had performed during screening. You will also have additional blood drawn (about 1-2 tablespoons each time) to check any tumor markers that were found to be increased in your blood during the screening tests.

In order to learn about the flow of blood to the tumor, non-routine functional CT scans will be performed at the end of Cycles 1 and 3. When possible, these scans will be performed at the same times as the routine CT scans.

Length of Study Treatment:

You may receive up to 12 cycles of study treatment, as long as you are benefitting. You will be taken off study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. RAD001 is not commercially available or FDA approved for this type of cancer. Avastin is commercially available and FDA approved for the treatment of advanced cancer of the colon and rectum. At this time, this drug combination is being used for research only.

Up to 36 patients will be enrolled in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed low or intermediate grade neuroendocrine carcinoma. Patients with neuroendocrine tumors associated with MEN1 syndrome will be eligible.
2. Patients must have at least one measurable site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) that has not been previously irradiated. If the patient has had previous radiation to the target lesion(s), there must be evidence of progression in the lesion(s) since the radiation.
3. Patients must have at least one lesion suitable for perfusion CT. The lesion should be greater than or equal to 3 cm in size in the cranial caudal direction.
4. Patients who are on a somatostatin analogue must be on a stable dose (no change in mg dose of long acting octreotide or lanreotide, changes in dosing interval of +/- 1 week is allowed) for 2 months prior to date of randomization.
5. Prior radiation therapy is permitted. A recovery period of at least 4 weeks after completion of radiotherapy is required prior to date of randomization.
6. Patients may have received prior interferon or cytotoxic chemotherapy. There are no limitations on the number of prior regimens. Patients who had no prior therapy are eligible. At least 28 days must have elapsed since last treatment.
7. Patients may have received prior therapy targeting c-kit, abl, Platelet Derived Growth Factor Receptor (PDGFR), or estimated glomerular filtration rate or epidermal growth factor receptor (EGFR) (imatinib, gefitinib, erlotinib, cetuximab).
8. Age >/= 18 years of age, because no dosing or adverse event data are currently available on the use of bevacizumab and everolimus in patients < 18 years of age.
9. Patients must have unresectable or metastatic disease.
10. Zubrod performance status of 0 or 1.
11. Patients must have adequate organ and marrow function as defined below: Leukocytes >/= 3,000/mcL; absolute neutrophil count >/=1,500/mcL; platelets >/=120,000 /mcL; total bilirubin </=1.5 times the institutional upper limit of normal (ULN); aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) </=3.0 times institutional ULN (</= 5 * ULN in patients with liver metastases); creatinine </= 2.0 OR, creatinine clearance >/= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
12. Patients not on anticoagulation must have Prothrombin time (PT)/partial thromboplastin time (PTT) within 1.2 * the upper limit of normal.
13. Patients on full-dose anticoagulation (warfarin or low molecular weight heparin) are eligible provided that both of the following criteria are met: The patient has an in-range INR (between 2 and 3) on a stable (no change in the prior 2 weeks) dose of oral anticoagulant or on a stable (no change in the prior 2 weeks) dose of low molecular weight heparin. The patient has no active bleeding or known pathological condition that carries a high risk of bleeding such as varices.
14. Patients must have resting blood pressure (BP) no greater than 140 mmHg (systolic) or 90 mmHg (diastolic) for eligibility. Initiation or adjustment of BP medication is permitted prior to date of randomization.
15. Women of child-bearing potential must have a negative urine pregnancy test within 7 days prior to date of randomization. Women who have had menses within the past 2 years, who have not had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy are considered to be of child-bearing potential.
16. Ability to understand and the willingness to sign a written informed consent document and ability to comply with study and/or follow-up procedures.
17. Men and women of reproductive potential must use effective means of contraception. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Barrier method of contraception is required during the study. Contraception should continue for 6 months after the last dose of bevacizumab.

Exclusion Criteria:

1. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
2. Prior treatment with a mTOR inhibitor or bevacizumab.
3. Chronic treatment with systemic steroids or another immunosuppressive agent.
4. A known history of immunocompromise, including a positive HIV test. An HIV test will not be required; however, previous medical history will be reviewed.
5. Inadequately controlled hypertension (defined as systolic blood pressure >140 and/or diastolic blood pressure > 90 mmHg on antihypertensive medications).
6. Any prior history of hypertensive crisis or hypertensive encephalopathy.
7. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
8. History of myocardial infarction or unstable angina within 6 months prior to date of randomization.
9. History of stroke or transient ischemic attack within 6 months prior to date of randomization.
10. Known history of brain or leptomeningeal metastases.
11. Significant vascular disease (e.g., aortic aneurysm, aortic dissection).
12. Symptomatic peripheral vascular disease.
13. Evidence of bleeding diathesis or coagulopathy.
14. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to date of randomization or anticipation of need for major surgical procedure during the course of the study.
15. Minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to date of randomization.
16. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to date of randomization.
17. Serious, non-healing wound, ulcer, or bone fracture.
18. Proteinuria at screening as demonstrated by either: urine protein:creatinine (UPC) ratio >/= 1.0 at screening, OR, Urinalysis for proteinuria >/= 2+ (patients discovered to have>/= 2+ proteinuria on urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
19. Known hypersensitivity to any component of bevacizumab.
20. Pregnant or lactating. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Yao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yao JC, Phan AT, Hess K, Fogelman D, Jacobs C, Dagohoy C, Leary C, Xie K, Ng CS. Perfusion computed tomography as functional biomarker in randomized run-in study of bevacizumab and everolimus in well-differentiated neuroendocrine tumors. Pancreas. 2015 Mar;44(2):190-7. doi: 10.1097/MPA.0000000000000255. PMID 25426617
- See also: UT MD Anderson Cancer Center website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited starting on January 17, 2008 to February 26, 2010. All recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: A total of forty-one (41) participants were enrolled in the trial but two (2) participants were not eligible due to screen failure, therefore, they were not included in the group assignments.
Groups:
- Avastin: Cycle 1: (First 3 weeks of study) - Avastin 15 mg/kg intravenous (IV), Cycle 2: Avastin 15 mg/kg IV every 3 weeks, RAD001 10 mg orally daily for 3 weeks
- RAD001: Cycle 1: (First 3 weeks of study) - RAD001 10 mg orally daily for 21 Days, Cycle 2: Avastin 15 mg/kg IV every 3 weeks, RAD001 10 mg orally daily for 3 weeks
Period: Overall Study
Arm/Group | Avastin | RAD001
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avastin | RAD001 | Total
Number analyzed (Participants) | 19 | 20 | 39
Age Continuous [Median (Full Range); unit: years] | 57 [22 to 81] | 60 [33 to 74] | 59 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Net Change Relative to Baseline in Tumor Blood Flow
Description: Tumor blood flow (ml/min/100gm) determined by functional computed tomography (CT). Functional computed tomography (CT) at baseline, after first and third cycles (21 day cycles). Change (percentage) calculated as tumor blood flow measured at baseline compared to tumor blood flow measurement taken at end of Cycle 1, week 3 (21 days), and again at end of Cycle 3, Week 9 (63 days).
Time Frame: Baseline to end of Cycle 3 (63 days)
Measure: Mean (Standard Deviation); unit: ml/min/100gm
Groups:
- Avastin: Cycle 1 (First 3 weeks of study) - Avastin 15 mg/kg intravenous (IV) or RAD001 10 mg orally daily for 21 Days, Cycle 2: Avastin 15 mg/kg IV every 3 weeks, RAD001 10 mg orally daily for 3 weeks
Arm/Group | Avastin | RAD001
Number analyzed (Participants) | 19 | 20
ml/min/100gm
  Baseline to Week 3 | -0.44 (0.32) [73.2 to 40.98] | -0.12 (08.16) [66.89 to 58.73]
  Baseline to Week 9 | -0.60 (0.44) [73.2 to 29.07] | -0.40 (0.27) [66.89 to 40.15]

ADVERSE EVENTS:
Time Frame: 2 years and 1 month
Description: Adverse Events reported as whole participant group regardless of the agent order received since all patients received both RAD001 and Avastin after one cycle (3 week) of receiving either RAD001 or Avastin per randomization.
Groups:
- Avastin + RAD001: One agent (RAD001 or Avastin) then adding the second agent (Avastin or RAD001): Avastin 15 mg/kg intravenous (IV) every 3 weeks + RAD001 10 mg orally daily for 21 Days
Arm/Group | Avastin + RAD001
Serious Adverse Events (participants affected / at risk) | 35/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin + RAD001 (N=39)
ALT ELEVATION (Metabolism and nutrition disorders) | 2
ANEMIA (Blood and lymphatic system disorders) | 2
AST ELEVATION (Metabolism and nutrition disorders) | 3
FATIGUE (General disorders) | 3
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4
INFECTION (Infections and infestations) | 3
NAUSEA (Gastrointestinal disorders) | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 5
PROTEINURIA (Metabolism and nutrition disorders) | 5
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2
VOMITING (Gastrointestinal disorders) | 2
WEIGHT LOSS (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin + RAD001 (N=39)
ALT ELEVATION (Metabolism and nutrition disorders) | 5
ANEMIA (Blood and lymphatic system disorders) | 13
ANOREXIA (Gastrointestinal disorders) | 14
AST ELEVATION (Metabolism and nutrition disorders) | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 7
DIARRHEA (Gastrointestinal disorders) | 19
DIZZINESS (General disorders) | 7
DYSGEUSIA (Nervous system disorders) | 5
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 9
EDEMA (General disorders) | 18
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 25
FATIGUE (General disorders) | 24
FEVER (General disorders) | 9
FLATULENCE (Gastrointestinal disorders) | 5
HEADACHE (Nervous system disorders) | 11
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 17
HYPERTENSION (Cardiac disorders) | 20
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 20
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 6
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 6
INFECTION (Infections and infestations) | 22
INSOMNIA (General disorders) | 6
MUCOSITIS (Gastrointestinal disorders) | 24
NAIL CHANGE (Gastrointestinal disorders) | 9
NAUSEA (Gastrointestinal disorders) | 17
NEUTROPENIA (Blood and lymphatic system disorders) | 7
PERIPHERAL NEUROPATHY (Musculoskeletal and connective tissue disorders) | 7
PROTEINURIA (Metabolism and nutrition disorders) | 17
SKIN RASH (Skin and subcutaneous tissue disorders) | 6
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8
VOMITING (Gastrointestinal disorders) | 11
WEIGHT LOSS (Gastrointestinal disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No